CLINICAL TRIAL: NCT03240159
Title: Long Antagonist Protocol for IVF: a Proof of Concept for a Single Luteal GnRH- Antagonist Protocol
Brief Title: Long Antagonist Protocol for IVF With Single Luteal Dose of Degarelix
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assisting Nature (Other)
Responsible Party: Principal Investigator, Papanikolaou Evaggelos, Papanikolaou Evaggelos, MD, PhD, Assisting Nature
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Degarelix-AN003
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pregnancy, Ovarian
MeSH Terms: conditions — Pregnancy, Ovarian | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Deg-24mg (Active Comparator): Single dose of Degarelix 24mg, on day 24th of previous luteal face cycle. On day 2 of the cycle: will be measured: LH levels, estradiol levels, and FSH levels.
  ON day 1 of the stimulation (depending day of the cycle): will be measured: LH levels, estradiol levels, and FSH levels.
  On day 6 of the stimulation( depending day of the cycle):will be measured: LH levels, estradiol levels, and FSH levels.
  On day 8 of the stimulation( depending day of the cycle):will be measured: LH levels, estradiol levels, and FSH levels.
  On day 10 of the stimulation( depending day of the cycle):will be measured: LH levels, estradiol levels, and FSH levels.
  Interventions: Drug: Degarelix
- Deg-16mg (Active Comparator): Single dose of Degarelix 16mg, on day 24th of previous luteal face cycle. On day 2 of the cycle: will be measured: LH levels, estradiol levels, and FSH levels.
  ON day 1 of the stimulation (depending day of the cycle): will be measured: LH levels, estradiol levels, and FSH levels.
  On day 6 of the stimulation( depending day of the cycle):will be measured: LH levels, estradiol levels, and FSH levels.
  On day 8 of the stimulation( depending day of the cycle):will be measured: LH levels, estradiol levels, and FSH levels.
  On day 10 of the stimulation( depending day of the cycle):will be measured: LH levels, estradiol levels, and FSH levels.
  Interventions: Drug: Degarelix
- Deg-12mg (Active Comparator): Single dose of Degarelix 12mg, on day 24th of previous luteal face cycle.On day 2 of the cycle: will be measured: LH levels, estradiol levels, and FSH levels.
  ON day 1 of the stimulation (depending day of the cycle): will be measured: LH levels, estradiol levels, and FSH levels.
  On day 6 of the stimulation( depending day of the cycle):will be measured: LH levels, estradiol levels, and FSH levels.
  On day 8 of the stimulation( depending day of the cycle):will be measured: LH levels, estradiol levels, and FSH levels.
  On day 10 of the stimulation( depending day of the cycle):will be measured: LH levels, estradiol levels, and FSH levels.
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Degarelix 24mg Degarelix 16mg Degarelix 12mg
  Active Comparator:
  Down regulation of LH, during exposing in three different doses of Degarelix

SUMMARY:
A prospective study of three different doses of Degarelix in late luteal phase of women undergoing ovarian stimulation for IVF

DETAILED DESCRIPTION:
A prospective study of three different doses of Degarelix in late luteal phase of women undergoing ovarian stimulation for IVF:Single dose of Degarelix 24mg, 16mg and 12 mg, on day 24th of previous luteal face cycle. On day 2 of the cycle: will be measured: LH levels, estradiol levels, and FSH levels.

ON day 1 of the stimulation (depending day of the cycle): will be measured: LH levels, estradiol levels, and FSH levels.

On day 6 of the stimulation( depending day of the cycle):will be measured: LH levels, estradiol levels, and FSH levels.

On day 8 of the stimulation( depending day of the cycle):will be measured: LH levels, estradiol levels, and FSH levels.

On day 10 of the stimulation( depending day of the cycle):will be measured: LH levels, estradiol levels, and FSH levels.

ELIGIBILITY:
Inclusion Criteria:

* primary infertility
* age 18-39 years; body mass index (BMI) 18-29kg/m2;
* regular menstrual cycle of 26-35days,
* presumed to be ovulatory;
* early follicular- phase serum concentration of FSH within normal limits (1-12 IU/l).

Exclusion Criteria:

* women with diabetes and other metabolic disease
* women with heart disease, QT prolongation,heart failure
* elevated liver enzymes, liver failure, hepatitis
* women with inflammatory or autoimmune disease
* abnormal karyotype;
* polycystic ovarian syndrome,
* endometriosis stage III/IV;
* history of being a 'poor responder',
* defined as >20 days of gonadotrophin in a previous stimulation cycle, or any previous cancellation of a stimulation cycle due to limited follicular response, or development of less than 4 follicles 15 mm in a previous stimulation cycle; history of recurrent miscarriage; severe OHSS in a previous stimula- tion cycle or any contraindication for the use of gonadotrophins.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
LH levels | 4 days after injection of Degarelix
  Effectively down regulation of follicular LH levels (<14mIU/ml)/

CONTACTS AND LOCATIONS:
Overall Officials: Evaggelos Papanikolaou, MD, PhD, Principal Investigator — Assisting Nature; Robert Najdecki, MD, PhD, Principal Investigator — Assisting Nature
Locations (1):
- Assisting Nature, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Papanikolaou EG, Yarali H, Timotheou E, Grynberg M, Zafeiratis O, Tournaye H, Najdecki R. A Proof-of-Concept Clinical Trial of A Single Luteal Use of Long-Acting Gonadotropin-Releasing Hormone Antagonist Degarelix in Controlled Ovarian Stimulation for In Vitro Fertilization: Long Antagonist Protocol. Front Endocrinol (Lausanne). 2018 Mar 1;9:25. doi: 10.3389/fendo.2018.00025. eCollection 2018. PMID 29545772